CLINICAL TRIAL: NCT00001643
Title: Gene Analysis in Parkinson's Disease
Brief Title: Gene Analysis of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970173; 97-HG-0173
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-08-31

CONDITIONS: Parkinson's Disease
Keywords: Lewy Body; Mutation; Hereditary; Dominant; Sporadic; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
The purposes of this study are to identify the gene or genes responsible for an inherited form of Parkinson's disease and learn more about how the disease develops.

In Parkinson's disease, a deficiency of a brain chemical called dopamine impairs the function of the part of the brain that controls movement. As a result, patients may have difficulty moving or they may have uncontrolled movements of their hands and fingers. Parkinson's disease usually occurs sporadically, with no known cause. In a few families, however, the disease seems to be inherited through a gene mutation (change). There is a 50-50 chance that a parent with the mutated gene will pass it on to a child. Children who do inherit the abnormal gene may or may not go on to actually develop Parkinson's disease-the relative chance of this happening is not known.

Individuals 18 years of age and older from families in which Parkinson's disease appears to be inherited may be eligible for this study. Participants will have their medical records reviewed, provide a personal and family medical history (by telephone or in person), and have a small blood sample (2 tablespoons) taken for genetic studies. The total time required for the study is about 1 to 2 hours.

Participants are encouraged to meet with a NIH investigator or with a genetics specialist in their local area before testing to talk about the possible implications for themselves and their families of the test results....

DETAILED DESCRIPTION:
Mutational analysis in patients with Parkinson's disease and a positive family history will be undertaken in an effort to identify and better understand the function of defective genes that cause Parkinson's disease in these individuals. DNA from these individuals is an important resource for screening candidate genes for mutations, for confirming that genes identified by other approaches are altered in patients, and for defining the mutational spectrum in these genes (genotype/phenotype correlation).

Unrelated, anonymous normal individuals will serve as controls for sequence comparisons. Information about genotypes will not be communicated back to the individuals as part of this study. While mutational analysis will continue, no further participants will be recruited to this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals over the age of 18 from families in which there are three or more individuals affected with Parkinson's disease (within three generations) and the proband was the only affected person available or willing to participate in the study

The diagnosis must be supported by accepted clinical criteria: tremor, bradykinesia, and responsiveness to L-DOPA.

PD may be associated with dementia. The study will lose power if individuals with mental impairment and PD are excluded. For this reason, decisionally-impaired individuals will be enrolled.

EXCLUSION CRITERIA:

No one under 18 will be enrolled because, with the exception of the rare autosomal recessive PD due to parkin mutations, PD does not affect minors. Study design does not involve testing fetuses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 1997-08-29; Primary Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Polymeropoulos MH, Lavedan C, Leroy E, Ide SE, Dehejia A, Dutra A, Pike B, Root H, Rubenstein J, Boyer R, Stenroos ES, Chandrasekharappa S, Athanassiadou A, Papapetropoulos T, Johnson WG, Lazzarini AM, Duvoisin RC, Di Iorio G, Golbe LI, Nussbaum RL. Mutation in the alpha-synuclein gene identified in families with Parkinson's disease. Science. 1997 Jun 27;276(5321):2045-7. doi: 10.1126/science.276.5321.2045. PMID 9197268
- [Background] Polymeropoulos MH, Higgins JJ, Golbe LI, Johnson WG, Ide SE, Di Iorio G, Sanges G, Stenroos ES, Pho LT, Schaffer AA, Lazzarini AM, Nussbaum RL, Duvoisin RC. Mapping of a gene for Parkinson's disease to chromosome 4q21-q23. Science. 1996 Nov 15;274(5290):1197-9. doi: 10.1126/science.274.5290.1197. PMID 8895469
- [Background] Eldridge R, Ince SE. The low concordance rate for Parkinson's disease in twins: a possible explanation. Neurology. 1984 Oct;34(10):1354-6. doi: 10.1212/wnl.34.10.1354. No abstract available. PMID 6541307